CLINICAL TRIAL: NCT03148860
Title: Impact of Concomitant Methotrexate on Efficacy, Safety and Adherence of Ustekinumab-treatment in Patients With Active Psoriasis Arthritis
Brief Title: Impact of Concomitant MTX on Efficacy, Safety and Adherence of Ustekinumab-treatment in Patients With Active PsA
Acronym: MUST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Frank Behrens (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Dr. Frank Behrens, Coordinating Investigator and representative of sponsor, Fraunhofer Institute for Translational Medicine and Pharmacology ITMP
Organization: Fraunhofer Institute for Translational Medicine and Pharmacology ITMP (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TMP-1115_01
Record Dates: First submitted 2017-04-04; First posted 2017-05-11 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; Ustekinumab; Methotrexate; DAS28
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Methotrexate; Ustekinumab

STUDY DESIGN:
Intervention Model Description: randomised, placebo-controlled, double-blind, multicenter study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Methotrexate tablets will be encapsulated equal to Placebo to ensure blinding. Ustekinumab will be open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Methotrexate naive - Ustekinumab and Methotrexate (Active Comparator): Methotrexate naive subjects will be randomised to receive Methotrexate or Placebo, Ustekinumab will be given open-label
  Interventions: Drug: Methotrexate; Drug: Ustekinumab
- Methotrexate naive - Ustekinumab and Placebo to Methotrexate (Placebo Comparator): Methotrexate naive subjects will be randomised to receive Methotrexate or Placebo, Ustekinumab will be given open-label
  Interventions: Drug: Ustekinumab; Other: Placebo
- Methotrexate pre-treated subjects-Ustekinumab and Methotrexate (Active Comparator): subjects pretreated with Methotrexate will be randomised to receive Methotrexate or Placebo, Ustekinumab will be given open-label
  Interventions: Drug: Methotrexate; Drug: Ustekinumab
- Methotrexate pre-treated subjects-Ustekinumab and PLC (Placebo Comparator): subjects pretreated with Methotrexate will be randomised to receive Methotrexate or Placebo, Ustekinumab will be given open-label
  Interventions: Drug: Ustekinumab; Other: Placebo

INTERVENTIONS:
Drug: Methotrexate — subjects will receive once weekly 15 mg (3 capsules) MTX
  Arms: Methotrexate naive - Ustekinumab and Methotrexate; Methotrexate pre-treated subjects-Ustekinumab and Methotrexate
Drug: Ustekinumab — subject will receive Ustekinumab open-label over a treatment period of 52 weeks
  Other Names: Stelara
Other: Placebo — subjects will receive once weekly 3 capsules PLC to MTX
  Arms: Methotrexate naive - Ustekinumab and Placebo to Methotrexate; Methotrexate pre-treated subjects-Ustekinumab and PLC

SUMMARY:
Methotrexate (MTX) co-medication can improve the therapeutic effect of biological therapies (e.g. Tumor necrosis factor (TNF) -inhibitors) in rheumatoid arthritis (RA), but its role in Psoriatic Arthritis (PsA) remains unclear.

No data from Randomized Clinical Trials (RCTs) are available to address the questions whether add-on of MTX to UST monotherapy, or a withdrawal of continuous MTX therapy in patients with newly initiated Ustekinumab (UST) treatment or simultaneously induction of MTX with UST in naive active PsA-patients will influence outcome measurements.

So, the purpose of the study is to analyse the effects of blinded MTX-co-medication on outcome in patients treated with UST: Non-inferiority at week 24 of UST monotherapy compared to add-on to MTX in patients with active PsA and at least 12 weeks of MTX treatment prior to screening or who are actually not treated with MTX and do not have prior inadequate response to MTX-treatment for PsA will be demonstrated.

DETAILED DESCRIPTION:
Methotrexate (MTX) co-medication can improve the therapeutic effect of biological therapies (e.g. TNF-inhibitors) in rheumatoid arthritis (RA), but its role in Psoriatic Arthritis (PsA) remains unclear. Differences in phenotypical manifestations between PsA and RA might influence the impact of co-medication, treatment response and treatment adherence differently.

Independent from this data, the impact of use of MTX in Ustekinumab (UST) treated patients with active PsA remains unclear: No data from Randomized Clinical Trials (RCTs) are available to address the questions whether add-on of MTX to UST monotherapy, or the other way around, a withdrawal of continuous MTX therapy in patients with newly initiated UST treatment or simultaneously induction of MTX with UST in patients will influence outcome.

There is some evidence that MTX may contribute to improved treatment persistence with anti-TNF therapy, particularly when used in combination with infliximab, but there is very little data to support a benefit in effectiveness in patients receiving concomitant MTX.

Additionally, MTX may play a role in immunogenicity: In the PSUMMIT program the patients with concomitant MTX had lower anti-drug-antibody (ADA) rates than those on UST-monotherapy, although there was no effect on efficacy and safety.

Furthermore, methotrexate treatment manifestations such as dactylitis or enthesitis seems to be ineffective.

In this study, the effect of blinded MTX-co-medication on outcome in patients treated with UST will be analysed. Differences on efficacy, safety and treatment adherence will be calculated related to MTX use in four arms of the stratified, randomized placebo-controlled clinical trial which contains a study treatment period of 52 weeks. The primary endpoint, differences in DAS28 in the treatment groups, will be measured at week 24.

ELIGIBILITY:
Inclusion Criteria:

Patients with active psoriatic arthritis who are naïve to UST will be stratified to either without MTX-therapy or on MTX-treatment (dosage 15mg once weekly) for at least 12 weeks prior to screening.

* Active PsA is defined as TJC ≥4 and SJC ≥4 (68/66 joint count) and DAS28 ≥ 3,2 at screening
* PsA according to CASPAR criteria
* At least age of 18 years
* Presence of chest x-ray without signs of active or latent infection (esp. for tuberculosis) within the last 3 months
* Permitted pre-treatment with up to three biologic-agents, whereupon only one biologic agent must be withdrawn due to inadequate response.
* For MTX-naive patients: Previous use of NSAID
* Written informed consent obtained prior to the initiation of any protocol-required procedures
* Compliance to study procedures and study protocol Inclusion criteria related to MTX
* For the group on MTX: Patients must have stable MTX dosages of at least 15mg once weekly for at least 12 weeks prior to screening and stable MTX dosages of at 15mg once weekly for at least 4 weeks prior to screening
* Compliance of intake of MTX must be documented by treating physician
* For the group without MTX therapy: patients must be eligible for MTX treatment (according to SmPC) and have not failed prior MTX treatment for the treatment of PsA

Exclusion Criteria:

Exclusion criteria related to Investigational medicinal product (IMP):

* Previous use of UST or any other anti-IL23 agent
* according to SmPC

Exclusion criteria for the group without MTX:

- Inadequate Response to prior MTX-treatment for Psoriatic Arthritis

Exclusion criteria related to general health:

* previous B-cell depleting therapy
* Patients with other chronic inflammatory articular disease or systemic autoimmune disease with musculoskeletal symptoms
* Patients with active Tb
* Patients with latent Tb, measured by Interferon gamma release assay, that are not pre-treated for at least 1 months and planned to be treated 9 months in total with INH once a day according to local guidelines
* Any active infection, a history of recurrent clinically significant infection, a history of recurrent bacterial infections with encapsulated organisms
* Primary or secondary immunodeficiency
* History of cancer with curative treatment not longer than 5 years ago except basal-cell carcinoma of the skin that had been excised
* Evidence of significant uncontrolled concomitant diseases or serious and/or uncontrolled diseases that are likely to interfere with the evaluation of the patient's safety and of the study outcome
* History of a severe psychological illness or condition
* Known hypersensitivity to any component of the product
* Women lactating, pregnant, nursing or of childbearing potential with a positive pregnancy test
* Males or females of reproductive potential not willing to use effective contraception (e.g. contraceptive pill, IUD, physical barrier)
* Alcohol, drug or chemical abuse Exclusion criteria related to prior treatments
* Previous DMARD therapy other than MTX at least for the last 28 days prior screening due to washout time of different DMARD therapies (including Leflunomide etc.)
* Previous immunosuppressive biologic therapy at least for the last
* 4 weeks prior to screening for Enbrel® (etanercept) - with a terminal half-life of 102 ± 30 hours (s.c. route)
* 10 weeks prior to screening for Humira® (adalimumab) - with a terminal half-life of 10-20 days (average 2 weeks) (s.c. route)
* 10 weeks prior to screening for Simponi® (golimumab) - with a terminal half-life of 11-14 days
* 10 weeks prior to screening for Cimzia® (certolizumab) - with a terminal half-life of approx. 14 days
* 8 weeks prior to screening for Remicade® (infliximab) - with a terminal half-life of 8.0-9.5 days (i.v. infusion)
* 60 days prior to screening due to washout time of other immunosuppressive biologic therapies
* current participation in another interventional clinical trial

Exclusion criteria related to laboratory:

* Haemoglobin < 8.5 g / dl
* Neutrophil counts < 1.500 / μl
* Platelet count < 75.000 / μl
* Lower than 1 x 1000 / μl lymphopenia for more than three months prior to inclusion.
* Serum creatinine > 1.4 mg / dl for women or 1.6 mg / dl for men
* AST or ALT > 2.5 time upper limit of norm

Exclusion criteria related to formal aspects:

- Underage or incapable patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Assessment of mean values of DAS28 at week 24 | week 24
  To demonstrate non-inferiority of mean values of DAS28 at week 24 of UST monotherapy compared to add-on to MTX with stratification according to patients on or without MTX before randomization.

SECONDARY OUTCOMES:
Assessment of mean DAS28 at week 52 | week 52
  The Disease Activity Score (DAS) consists of SJC and TJC measurements, the erythrocyte sedimentation rate (or CRP) and the subject's global assessment of disease activity.
Assessment of DAS28 | week 4
  The Disease Activity Score (DAS) consists of SJC and TJC measurements, the erythrocyte sedimentation rate (or CRP) and the subject's global assessment of disease activity.
Assessment of DAS28 | week 16
  The Disease Activity Score (DAS) consists of SJC and TJC measurements, the erythrocyte sedimentation rate (or CRP) and the subject's global assessment of disease activity.
Assessment of DAS28 | week 24
  The Disease Activity Score (DAS) consists of SJC and TJC measurements, the erythrocyte sedimentation rate (or CRP) and the subject's global assessment of disease activity.
Assessment of DAS28 | week 40
  The Disease Activity Score (DAS) consists of SJC and TJC measurements, the erythrocyte sedimentation rate (or CRP) and the subject's global assessment of disease activity.
Assessment of DAS28 | week 52
  The Disease Activity Score (DAS) consists of SJC and TJC measurements, the erythrocyte sedimentation rate (or CRP) and the subject's global assessment of disease activity.
change in DAS28 | baseline to week 4
  The Disease Activity Score (DAS) consists of SJC and TJC measurements, the erythrocyte sedimentation rate (or CRP) and the subject's global assessment of disease activity.
change in DAS28 | baseline to week 16
  The Disease Activity Score (DAS) consists of SJC and TJC measurements, the erythrocyte sedimentation rate (or CRP) and the subject's global assessment of disease activity.
change in DAS28 | baseline to week 24
  The Disease Activity Score (DAS) consists of SJC and TJC measurements, the erythrocyte sedimentation rate (or CRP) and the subject's global assessment of disease activity.
change in DAS28 | baseline to week 40
  The Disease Activity Score (DAS) consists of SJC and TJC measurements, the erythrocyte sedimentation rate (or CRP) and the subject's global assessment of disease activity.
change in DAS28 | baseline to week 52
  The Disease Activity Score (DAS) consists of SJC and TJC measurements, the erythrocyte sedimentation rate (or CRP) and the subject's global assessment of disease activity.
DAS28-ESR remission | week 4
DAS28-ESR remission | week 16
DAS28-ESR remission | week 24
DAS28-ESR remission | week 40
DAS28-ESR remission | week 52
Assessment of Tender joint count/Swollen joint count (TJC/SJC) (68/66) | week 4
  Tender and swollen joint will be assessed and counted by trained personel
Assessment of TJC/SJC (68/66) | week 16
  Tender and swollen joint will be assessed and counted by trained personel
Assessment of TJC/SJC (68/66) | week 24
  Tender and swollen joint will be assessed and counted by trained personel
Assessment of TJC/SJC (68/66) | week 40
  Tender and swollen joint will be assessed and counted by trained personel
Assessment of TJC/SJC (68/66) | week 52
  Tender and swollen joint will be assessed and counted by trained personel
ACR (20/50/70) response | week 4
  Portion of Patient that reach 20%, 50% or 70% improvement in ACR score consisting of SJC and TJC measurements, subject's assessment of pain, subject's global assessment of disease activity, physician's global assessment of disease activity, HAQ and measurements of erythrocyte sedimentation rate and CRP
ACR (20/50/70) response | week 16
  Portion of Patient that reach 20%, 50% or 70% improvement in ACR score consisting of SJC and TJC measurements, subject's assessment of pain, subject's global assessment of disease activity, physician's global assessment of disease activity, HAQ and measurements of erythrocyte sedimentation rate and CRP
ACR (20/50/70) response | week 24
  Portion of Patient that reach 20%, 50% or 70% improvement in ACR score consisting of SJC and TJC measurements, subject's assessment of pain, subject's global assessment of disease activity, physician's global assessment of disease activity, HAQ and measurements of erythrocyte sedimentation rate and CRP
ACR (20/50/70) response | week 40
  Portion of Patient that reach 20%, 50% or 70% improvement in ACR score consisting of SJC and TJC measurements, subject's assessment of pain, subject's global assessment of disease activity, physician's global assessment of disease activity, HAQ and measurements of erythrocyte sedimentation rate and CRP
ACR (20/50/70) response | week 52
  Portion of Patient that reach 20%, 50% or 70% improvement in ACR score consisting of SJC and TJC measurements, subject's assessment of pain, subject's global assessment of disease activity, physician's global assessment of disease activity, HAQ and measurements of erythrocyte sedimentation rate and CRP
Change in ACR core set | baseline to week 4
  Changes in SJC, TJC, HAQ, patient's and physician's global assessment, pain, CRP and ESR will be described
Change in ACR core set | baseline to week 16
  Changes in SJC, TJC, HAQ, patient's and physician's global assessment, pain, CRP and ESR will be described
Change in ACR core set | baseline to week 24
  Changes in SJC, TJC, HAQ, patient's and physician's global assessment, pain, CRP and ESR will be described
Change in ACR core set | baseline to week 40
  Changes in SJC, TJC, HAQ, patient's and physician's global assessment, pain, CRP and ESR will be described
Change in ACR core set | baseline to week 52
  Changes in SJC, TJC, HAQ, patient's and physician's global assessment, pain, CRP and ESR will be described
Assessment of PASI | week 4
  The Psoriasis Area and Severity Index (PASI) is used for evaluation of severity and extend of skin involvement of the included patients
Assessment of BASDAI | week 4
  The Bath ankylosing spondylitis disease activity index will be performed for those patients who have radiological findings suspect for axial involvement
Assessment of BSA | week 4
  The body surface area will be evaluated to measure the extend of Psoriasis in the included PsA patients.
Assessment of BASDAI | week 16
  The Bath ankylosing spondylitis disease activity index will be performed for those patients who have radiological findings suspect for axial involvement
Assessment of PASI | week 16
  The Psoriasis Area and Severity Index (PASI) is used for evaluation of severity and extend of skin involvement of the included patients
Assessment of BSA | week 16
  The body surface area will be evaluated to measure the extend of Psoriasis in the included PsA patients.
Assessment of BASDAI | week 24
  The Bath ankylosing spondylitis disease activity index will be performed for those patients who have radiological findings suspect for axial involvement
Assessment of PASI | week 24
  The Psoriasis Area and Severity Index (PASI) is used for evaluation of severity and extend of skin involvement of the included patients
Assessment of BSA | week 24
  The body surface area will be evaluated to measure the extend of Psoriasis in the included PsA patients.
Assessment of PASI | week 40
  The Psoriasis Area and Severity Index (PASI) is used for evaluation of severity and extend of skin involvement of the included patients
Assessment of BSA | week 40
  The body surface area will be evaluated to measure the extend of Psoriasis in the included PsA patients.
Assessment of BASDAI | week 40
  The Bath ankylosing spondylitis disease activity index will be performed for those patients who have radiological findings suspect for axial involvement
Assessment of PASI | week 52
  The Psoriasis Area and Severity Index (PASI) is used for evaluation of severity and extend of skin involvement of the included patients
Assessment of BSA | week 52
  The body surface area will be evaluated to measure the extend of Psoriasis in the included PsA patients.
Assessment of BASDAI | week 52
  The Bath ankylosing spondylitis disease activity index will be performed for those patients who have radiological findings suspect for axial involvement
Treatment adherence measured by patient diary | through treatment period; normally 52 weeks
  Compliance with treatment will be determined by patient diary
Compliance measured by questionnaire CQR5 | through treatment period; normally 52 weeks
  The CQR5 consists of 5 questions addressing information on treatment compliance of the patient.
Quality of life measured by HAQ | week 4
  Stanford Health Assessment Questionnaire disability index is a patient reported questionnaire specific for RA
Quality of life measured by EQ5D | week 4
  EQ5D is a standardised instrument for use as a measure of health outcome
Quality of life measured by DLQI | week 4
  The Dermatology Life Quality Index is a 10-question validated questionnaire.
Quality of life measured by EQ5D | week 16
  EQ5D is a standardised instrument for use as a measure of health outcome
Quality of life measured by HAQ | week 16
  Stanford Health Assessment Questionnaire disability index is a patient reported questionnaire specific for RA
Quality of life measured by DLQI | week 16
  The Dermatology Life Quality Index is a 10-question validated questionnaire.
Quality of life measured by DLQI | week 24
  The Dermatology Life Quality Index is a 10-question validated questionnaire.
Quality of life measured by EQ5D | week 24
  EQ5D is a standardised instrument for use as a measure of health outcome
Quality of life measured by HAQ, | week 24
  Stanford Health Assessment Questionnaire disability index is a patient reported questionnaire specific for RA
Quality of life measured by HAQ | week 40
  Stanford Health Assessment Questionnaire disability index is a patient reported questionnaire specific for RA
Quality of life measured by EQ5D | week 40
  EQ5D is a standardised instrument for use as a measure of health outcome
Quality of life measured by DLQI | week 40
  The Dermatology Life Quality Index is a 10-question validated questionnaire.
Quality of life measured by HAQ | week 52
  Stanford Health Assessment Questionnaire disability index is a patient reported questionnaire specific for RA
Quality of life measured by EQ5D | week 52
  EQ5D is a standardised instrument for use as a measure of health outcome
Quality of life measured by DLQI | week 52
  The Dermatology Life Quality Index is a 10-question validated questionnaire.
Assessment of Change in Dactylitis | week 4, 16, 24, 40 and week 52
  Functional assessment: Change in number and severity of digits involved) involved
Assessment of Change in Enthesitis (LEI) | week 4, 16, 24, 40 and week 52
  functional outcome
Assessment of mtNAPSI | week 4, 16, 24, 40 and week 52
  The modified target Nail Psoriasis Severity Index is used for evaluation of nail involvement in patients
Ultrasound (US) assessment of joints and enthesis according to PASON22 | Week 4, 24 and week 52
  selected sites only
Frequency and seriousness of adverse events as reported and documented in Case report form | each study visit (week 0 to week 52)
  Documentation of the occurence, frequency and seriousness of adverse events as reported and documented in Case report form

CONTACTS AND LOCATIONS:
Overall Officials: Frank Behrens, MD, Principal Investigator — Fraunhofer IME
Locations (1):
- CIRI, Frankfurt am Main, Hessia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koehm M, Rossmanith T, Foldenauer AC, Herrmann E, Brandt-Jurgens J, Burmester GR, Kellner H, Kiltz U, Kofler DM, Rech J, Mojtahed-Poor S, Jonetzko C, Burkhardt H, Behrens F; MUST Investigator Group. Methotrexate plus ustekinumab versus ustekinumab monotherapy in patients with active psoriatic arthritis (MUST): a randomised, multicentre, placebo-controlled, phase 3b, non-inferiority trial. Lancet Rheumatol. 2023 Jan;5(1):e14-e23. doi: 10.1016/S2665-9913(22)00329-0. PMID 38251504
- [Derived] Mojtahed Poor S, Henke M, Ulshofer T, Kohm M, Behrens F, Burkhardt H, Schiffmann S. The role of antidrug antibodies in ustekinumab therapy and the impact of methotrexate. Rheumatology (Oxford). 2023 Dec 1;62(12):3993-3999. doi: 10.1093/rheumatology/kead177. PMID 37079726